CLINICAL TRIAL: NCT00003372
Title: A Phase II Study of Topotecan in Patients With Anaplastic Oligodendroglioma or Anaplastic Mixed Oligoastrocytoma
Brief Title: Topotecan in Treating Patients With Recurrent Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I109; CAN-NCIC-IND109 (Other: PDQ); CDR0000066362 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-06-09 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult anaplastic oligodendroglioma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Oligodendroglioma; Glioma | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of topotecan in treating patients with recurrent brain tumor.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of topotecan in patients with recurrent anaplastic oligodendroglioma or anaplastic mixed oligoastrocytoma. II. Determine the qualitative and quantitative toxicity of topotecan in this patient population on this schedule.

OUTLINE: This is a multicenter study. Patients receive intravenous topotecan over 30 minutes daily for 5 days every 3 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients will be followed every 3 months until death.

PROJECTED ACCRUAL: Up to 30 evaluable patients will be accrued within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent anaplastic oligodendroglioma or anaplastic mixed oligoastrocytoma following primary surgery and radiation therapy Tumors for anaplastic mixed oligoastrocytoma must contain at least 25% oligodendroglial elements Tumors must be clinically aggressive for patients with only 1 anaplastic feature Prior low grade oligodendrogliomas or oligoastrocytomas undergoing repeat biopsy following clinical or radiological progression are eligible Bidimensionally measurable and progressive lesions by CT or MRI

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-3 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Not specified Renal: Creatinine normal Other: Not pregnant or nursing Fertile patients must use effective contraception No prior malignancies except curatively treated carcinoma in situ of the cervix or nonmelanoma skin cancer No other serious illness or medical condition No active uncontrolled infection No history of neurologic or psychiatric disorder

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 6 weeks since chemotherapy No more than 1 prior chemotherapy regimen No prior camptothecin derivatives Endocrine therapy: At least 2 weeks on stable steroid therapy, if necessary Radiotherapy: At least 2 months since prior radiotherapy No prior radiation therapy for recurrent disease Surgery: At least 6 weeks since prior surgery (except biopsy only) Prior surgery for recurrent disease allowed (including stereotactic biopsy or partial resection) Other: No concurrent experimental drugs or anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 1997-12-08 (Actual); Primary Completion 2000-10-05 (Actual); Study Completion 2009-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Belanger, MD, Study Chair — CHUM - Hotel Dieu Hospital
Locations (11):
- Canada (11):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre - Civic Campus, Ottawa, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Belanger K, MacDonald D, Cairncross G, Gertler S, Forsyth P, Burdette-Radoux S, Bergeron J, Soulieres D, Ludwin S, Wainman N, Eisenhauer E. A phase II study of topotecan in patients with anaplastic oligodendroglioma or anaplastic mixed oligoastrocytoma. Invest New Drugs. 2003 Nov;21(4):473-80. doi: 10.1023/a:1026211620793. PMID 14586216